CLINICAL TRIAL: NCT00686257
Title: Evaluation Of The Total Face Mask For Emergency Application In Acute Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-6060
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-05

CONDITIONS: Acute Respiratory Insufficiency
Keywords: acute respiratory insufficiency; noninvasive ventilation; oronasal face mask; total face mask

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients receiving NPPV by the 'Total Face Mask'
  Interventions: Device: Total face mask (interface for NPPV)
- 2 (Active Comparator): Patients receiving NPPV by 'standard oronasal mask'
  Interventions: Device: Comfort full or RT040 oronasal mask (interface for NPPV)

INTERVENTIONS:
Device: Total face mask (interface for NPPV) — NPPV is applied by this mask, as long as NPPV is received.
  Other Names: cephalic mask
  Arms: 1
Device: Comfort full or RT040 oronasal mask (interface for NPPV) — NPPV is applied by one of these masks (Comfort full or RT040 masks used at Rhode Island Hospital and Tufts Medical Center respectively), as long as NPPV is received.
  Other Names: Full face mask
  Arms: 2

SUMMARY:
The purpose of this study is to compare the Total Face Mask™ (Respironics, Inc., Pittsburgh, PA) (covering whole face) and the standard oronasal facemask (covering nose and mouth) for the emergency treatment of patients with acute respiratory failure with the machine blowing air into the mask placed on the face (noninvasive positive pressure ventilation) (NPPV).

DETAILED DESCRIPTION:
Despite its demonstrated efficacy in treating selected patients with acute respiratory failure, the application of NPPV is still plagued by a substantial failure rate, ranging from below 10% to above 40%. Mask intolerance ranks as one of the most common causes of failure. This is related to ill-fitting masks, mask discomfort (despite a properly fitted mask), excessively tightened straps, excessive air leaks around the mask or through the mouth, and claustrophobia.

The most commonly used masks in the acute care setting are either oronasal masks that cover the nose and mouth, or nasal masks that cover the nose alone. Both mask types usually consist of clear plastic dome-shaped mask with a soft silicon gasket to create an air seal with the skin. While this approach is usually successful, it may lead to patient discomfort and/or an air leak secondary to the difficulty in creating an effective seal over the bridge of the nose and over mobile structures such as the mandible. The Total Face Mask ™ (Respironics, Inc., Pittsburgh, PA) uses a different approach to avoid some of these limitations. Considerably larger than a standard oronasal mask, it covers the entire face and creates an air seal using a silicon gasket around the parameter of the face. In this way, gasket pressure is more evenly distributed, and discomfort over the bridge of the nose or chin is eliminated, and air leaking reduced. In addition, because one mask size fits virtually all patients, the Total Face Mask ™ facilitates the fitting process and permits more rapid initiation of ventilatory assistance. Clinical experience to date suggests that claustrophobia is not a common problem with the Total Face Mask ™ despite its size, and that its contribution to dead space is comparable to that of most oronasal masks.

The following protocol aims to compare use of the Total Face Mask ™ to the Comfort Full oronasal mask (also by Respironics, Inc., Pittsburgh, PA)or RT040 oronasal mask (Fisher&Paykel Inc., Wellington, NZ) in the acute care setting for patients meeting standard indications for NPPV.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Either A or B

A. Clinical Criteria: Moderate to severe respiratory distress as evidenced by tachypnea, use of accessory muscles for breathing, or abdominal paradox.

B. Blood Gas and Physiologic Criteria: Gas exchange abnormalities including PaCO2>45 with a pH<7.35, or a PaO2/FiO2 ratio<200.

Exclusion Criteria:

* The need for immediate intubation
* Medical instability such as hypotensive shock, uncontrolled cardiac ischemia or arrythmias, unstable myocardial infarction, uncontrolled upper gastrointestinal bleeding
* Agitation or uncooperativeness, unresponsive to small doses of sedatives
* Excretions or inability to protect the airway
* Inability to fit the mask
* Facial trauma
* Upper airway obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aylin Ozsancak, MD, Study Chair — Research Fellow; Nicholas S. Hill, MD, Principal Investigator — Chair of Pulmonary, Critical Care and Sleep Division; Samy Sidhom, MD, MPH, Study Director — Clinical Fellow
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Result] Ozsancak A, Sidhom SS, Liesching TN, Howard W, Hill NS. Evaluation of the total face mask for noninvasive ventilation to treat acute respiratory failure. Chest. 2011 May;139(5):1034-1041. doi: 10.1378/chest.10-1905. Epub 2011 Feb 17. PMID 21330385

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Face Mask: Patients receiving NPPV by the 'Total Face Mask' or standard face mask controls
- Standard Face Mask Controls: Patients receiving NPPV by 'standard oronasal mask'
Period: Overall Study
Arm/Group | Total Face Mask | Standard Face Mask Controls
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Face Mask | Standard Face Mask Controls | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (15) | 62.6 (17) | 62.9 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Mask Comfort (as Determined by the Visual Analog Scores 1 Being Least, 10 Being Most)
Time Frame: During the first 3 hours of recruitment
Population: By power analysis
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Control: Received standard face mask
- Total Face Mask: Received Total Face Mask
Arm/Group | Control | Total Face Mask
Number analyzed (Participants) | 31 | 29
units on a scale | 3.2 (0.6) | 3.3 (0.7)

2. Primary Outcome: Time Required for Mask Placement
Time Frame: at the initiation of NPPV
Measure: Median (Inter-Quartile Range); unit: Minutes
Groups:
- Oronosal Mask: Standard oronosal mask
- Total Face Mask: Total Face Mask
Arm/Group | Oronosal Mask | Total Face Mask
Number analyzed (Participants) | 31 | 29
Minutes | 5 [2 to 8] | 3.5 [1.9 to 5]

3. Secondary Outcome: Early NIV Discontinuation Rate
Description: Defined as the inability of the patient to be maintained on NPPV using the assigned mask while there was still an indication for ventilatory support
Time Frame: During hospitalization period (after recruitment into the study)
Measure: Count of Participants; unit: Participants
Arm/Group | Oronosal Mask | Total Face Mask
Number analyzed (Participants) | 31 | 29
Participants | 12 | 16

4. Secondary Outcome: Deterioration Vital Signs
Time Frame: during the first 24 hours of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Oronosal Mask | Total Face Mask
Number analyzed (Participants) | 31 | 29
Participants | 7 | 3

5. Secondary Outcome: Deterioration in Gas Exchange
Time Frame: during the first 24 hours of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Total Face Mask
Number analyzed (Participants) | 31 | 29
Participants | 3 | 3

6. Secondary Outcome: Total Length of Time Requiring NIV
Time Frame: during hospitalization (after recruitment)
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Oronosal Mask | Total Face Mask
Number analyzed (Participants) | 31 | 29
Hours | 15.7 [4.0 to 49.8] | 6.05 [0.9 to 56.7]

7. Secondary Outcome: Length of Hospital Stay
Time Frame: during hospitalization (after recruitment)
Measure: Mean (Full Range); unit: Days
Arm/Group | Oronosal Mask | Total Face Mask
Number analyzed (Participants) | 31 | 29
Days | 19.2 [5 to 92] | 10.9 [1 to 77]

8. Secondary Outcome: In-hospital Mortality Rate
Time Frame: during hospitalization (after recruitment)
Measure: Count of Participants; unit: Participants
Arm/Group | Oronosal Mask | Total Face Mask
Number analyzed (Participants) | 31 | 29
Participants | 6 | 3

ADVERSE EVENTS:
Arm/Group | Total Face Mask | Standard Face Mask Controls
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 6/29 | 4/31
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Face Mask (N=29) | Standard Face Mask Controls (N=31)
Claustrophobia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) — Claustrophobia in 4 control patients and 6 Total Face mask patients

LIMITATIONS AND CAVEATS:
Could not blind subjects or investigators

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes